CLINICAL TRIAL: NCT01619293
Title: The Neuromarker S-100B in Patients With Subarachnoidal, Epidural, Subdural, and Intracerebral Hematoma, Edema Cerebri, and Concussion
Brief Title: The Neuromarker S-100B in Patients With Different Types of Intracranial Injury
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Harald Wolf, MD, Principal Investigator, Medical University of Vienna
Other Study IDs: Wolf-5
Record Dates: First submitted 2012-05-30; First posted 2012-06-14 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Traumatic Brain Injury; Trauma
Keywords: CCT; brain; trauma; injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 7ml of blood drawed from peripheral vein
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Epidural H.: patients with hematoma epidurale
- Subdural H.: patients with hematoma subdurale
- Subarachnoidal H.: patients with hematoma subarachnoidale
- Intracerebral H.: patients with hematoma intracerebrale
- E. cerebri: patients with edema cerebri
- Concussion: patients with concussion

SUMMARY:
Abstract:

The most widely studied neuro-markers in traumatic brain injury (TBI) are S100B and neurone specific enolase (NSE). S-100B is localized in astroglia. This marker is used to predict neuronal damage caused by traumatic brain injury. The investigators conduct a study to derive and validate the measurement of S-100B in serum of patients with different types traumatic brain injuries.

DETAILED DESCRIPTION:
The neuromarker S-100B is a well established tool for decision making in patients traumatic brain injury (TBI)in Europe. In many hospitals S-100B is used routinely as a part of a set of high- and medium risk factors aiding the decision to perform a cranial computed tomography (CCT) in patients with minor head injury (MHI). In patients with severe head injury Raabe et al. found a significant correlation between the S-100B levels and unfavourable outcome in patients with severe brain injury with serum levels higher than 0.50 μg/l measured 24h after injury. The average level of the neuromarker, compared with other studies. The study of Biberthaler et al. showed highest levels in patients with epidural hematomas, followed by subdural, subarachnoidal and intracerebral hematomas. On the contrary the average S-100B levels of patients with epidural hematomas featured in a study by Unden et al. published in 2005 displayed normal levels (<0.2 μg/L). They concluded that S-100B was unreliable as a marker for epidural hematomas.

Aim of the study Validation of S-100B in patients with intracerebral, epidural, subdural, and subarachnoidal hematoma, brain edema and concussion (Group 1-6), to find evidence which kind of injury leads to which level of elevation of the neuromarker measured in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* all patients with traumatic brain injury

Exclusion Criteria:

* patients without traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Level 1 trauma center
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
S100B LEVEL | 14 month
  S-100B level higher than 0.105 ug/L is held pathological

CONTACTS AND LOCATIONS:
Overall Officials: Harald Wolf, M.D., Principal Investigator — Dept. Trauma Surgery; Medical Univ. of Vienna, Austria
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Unden J, Bellner J, Astrand R, Romner B. Serum S100B levels in patients with epidural haematomas. Br J Neurosurg. 2005 Feb;19(1):43-5. doi: 10.1080/02688690500089381. PMID 16147582
- [Background] Biberthaler P, Linsenmeier U, Pfeifer KJ, Kroetz M, Mussack T, Kanz KG, Hoecherl EF, Jonas F, Marzi I, Leucht P, Jochum M, Mutschler W. Serum S-100B concentration provides additional information fot the indication of computed tomography in patients after minor head injury: a prospective multicenter study. Shock. 2006 May;25(5):446-53. doi: 10.1097/01.shk.0000209534.61058.35. PMID 16680008
- [Background] Mussack T, Kirchhoff C, Buhmann S, Biberthaler P, Ladurner R, Gippner-Steppert C, Mutschler W, Jochum M. Significance of Elecsys S100 immunoassay for real-time assessment of traumatic brain damage in multiple trauma patients. Clin Chem Lab Med. 2006;44(9):1140-5. doi: 10.1515/CCLM.2006.190. PMID 16958611